CLINICAL TRIAL: NCT00037830
Title: The Study of GM1 Ganglioside, A Potential New Parkinson's Disease Medication
Brief Title: GM1 Ganglioside Effects on Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS038681 (NIH); R01NS038681 (NIH)
Record Dates: First submitted 2002-05-22; First posted 2002-05-23 (Estimated); Results first posted 2012-08-09 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; PD; GM1 Ganglioside; Sygen
MeSH Terms: conditions — Parkinson Disease | interventions — G(M1) Ganglioside

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Early-Start Group (Active Comparator): Subjects were randomized to receive GM1 ganglioside for 24 weeks.
  Interventions: Drug: GM1 ganglioside
- Delayed-Start Group (Placebo Comparator): Subjects were randomized to receive placebo for 24 weeks.
  Interventions: Drug: Placebo
- Comparison Group (No Intervention): A separate group of Parkinson's disease patients who received standard of care were followed for one to two years to provide comparative information about natural disease progression. This comparison group was not compared statistically to the treatment groups since they were not randomized.

INTERVENTIONS:
Drug: GM1 ganglioside — 100 mg twice per day by subcutaneous injection
  Other Names: Sygen
  Arms: Early-Start Group
Drug: Placebo — Twice per day subcutaneous injection, equal volume as active drug
  Arms: Delayed-Start Group

SUMMARY:
The purpose of this trial is to examine the short term effects (24 Weeks) of GM1 on Parkinson's disease (PD) symptoms, as well as the effects of long-term treatment (120 Weeks) with GM1 on disease progression, and to examine the extent to which GM1 treatment influences the underlying disease process in PD.

DETAILED DESCRIPTION:
The study is designed to further examine the extent to which GM1 ganglioside can improve symptoms, delay disease progression, and, perhaps, partially restore damaged brain cells in PD patients. GM1 ganglioside is a chemical that is normally found in the brain and is a normal part of the outer covering or membrane of nerve cells. This study will compare the effectiveness of GM1 to standard PD treatment. In addition to studying clinical measures of motor and cognitive functioning, the investigators will use PET (positron emission tomography) scanning to image the brain and the dopamine nerve endings in a subgroup of patients. Patients with mild to moderate idiopathic PD will be divided into 2 groups. One group will receive GM1 for 24 weeks and the other will receive placebo. At the end of this 24 week period, all patients will enter into a 96 week treatment period in which all patients will receive GM1.

In parallel, a group of standard-of-care patients with mild to moderate PD will be monitored over a 1 to 2 year period to assess the natural progression of PD. These patients will receive the same clinical evaluations as the treatment group subjects but they will not receive the experimental medication.

ELIGIBILITY:
Inclusion criteria:

* Btwn ages of 39-85 yrs old.
* Females: at least 2 years post-menopausal; surgically sterile; or negative pregnancy test by quantitative serum ßHCG, & follow a reliable method of birth control for at least 2 months prior to entry, agree both to follow a reliable method of birth control, & to desist from breast feeding during, & for 1 month following, the study drug administration.
* Dx of idiopathic PD 6 months prior to screening. The diagnosis requires: the presence of at least 2 of the 4 cardinal clinical manifestations of the disease, tremor, rigidity, bradykinesia, and disturbances of posture or gait, & at least 1 must be rigidity or bradykinesia.
* Modified Hoehn and Yahr Staging between 1 and 3 as rated during an "off" period of at least 12 hours.
* Unified Parkinson's Disease Rating Scale motor component score between 10 and 40 as rated during an "off" period of at least 12 hours and a score of 6 or greater during "on" period.
* Antiparkinsonian treatments: stable treatment of l-dopa/carbidopa and/or dopamine agonist for at least 3 months prior to Screening.
* Mini Mental State Exam score > 25.
* Beck Depression Inventory score < 10.
* Signed informed consent.

Exclusion criteria:

* Abrupt onset of Parkinsonism.
* Failure of Parkinsonian symptoms to have responded to l-dopa.
* Motor symptoms (such as peak dose dyskinesias (UPDRS score > 3), & random on-off phenomenon, other than end-of-dose wearing-off, persistently fluctuating over a 6 month or longer period, in response to l-dopa.
* Hx of findings of any movement disorder other than idiopathic PD.
* A tremor score on the UPDRS motor scale of >5. Tremor score greater than 3 in an individual limb.
* High-dose vitamin E therapy (more than 1000 I.U./day) any time during the period starting 3 months prior baseline.
* Transient ischemic attack any time during the period starting 6 months prior baseline.
* Hx of 2 or more strokes. Hx of any stroke that resulted in motor deficit, movement disorder, ataxia, cognitive impairment, or a hemi-inattention syndrome. Any stroke with residua at the time of, or within 6 months preceding, study entry.
* Previous cerebral infarction, including lacunar infarction, in any area subserving motor function.
* Binswanger's disease or hx of hypertensive encephalopathy.
* Hx of encephalitis.
* Hx of extended exposure to any known neurotoxin that may cause parkinsonism, or chronic or sufficient use or consumption of any non-medicinal substance that could cause risk of developing a movement disorder or disturbance of posture or gait.
* Use of the following drugs within 6 months prior to screening: neuroleptics, metoclopramide, clozapine, flunarizine, alpha-methyldopa.
* Patients actively taking a medicine that is known to compete with the imaging agent for binding sites on the dopamine terminals.
* Hx of medication or drug use that may have caused atypical parkinsonism or history of Substance Use Disorder.
* Hx of a metabolic disorder that resulted or could have resulted in movement disorder or disturbance of posture or gait.
* Any disease or condition that resulted or could have resulted in a movement disorder or disturbance of posture or gait.
* Hx of intracranial hemorrhage, intracranial neoplasm, significant head trauma with loss of consciousness >24 hrs or other structural brain disease.
* Hx or clinical findings suggestive of progressive supranuclear palsy or multiple system atrophy.
* Acquired cognitive impairment reasonably possibly due to any cause other than idiopathic PD.
* Hx of a hereditary disorder associated with a movement disorder.
* Normal or low pressure hydrocephalus.
* Any ill-defined neuropathic disease, myelopathy, myopathy or other medical disorder or physical condition by history or clinical examination that could be expected to interfere with the diagnosis, treatment or assessment of PD, or with any of the study assessments.
* Hx of Guillain-Barré syndrome, chronic idiopathic polyneuropathy, or relapsing polyneuropathy.
* Hx of Axis I or Axis II major psychiatric disorder.
* Significant cardiac, pulmonary, hepatic, gastrointestinal, or renal disease.
* Any condition that could alter the distribution, accumulation, metabolism, or excretion of the study medication; or result in a life expectancy of less than 2 years.
* Any primarily non-neurologic medical condition with a significant risk of secondarily causing neurologic dysfunction.
* Myocardial infarction within 6 months prior to screening.
* Presence of any medical condition or laboratory test abnormality or use of any licit or illicit substance which could cause unwarranted risk from participation in the study or result in worsening in the patient's medical condition during participation in study. Presence of any of the following laboratory test abnormalities are unwarranted risk: serum transaminase greater than twice the upper limit of normal;serum creatinine greater than 2.0 mg/dl in a man or greater than 1.7 mg/dl in a woman.
* Hx of a life-threatening allergic or immune-mediated reaction.
* Previous use of any ganglioside preparation.
* Use of any experimental drug in the period starting 60 days before Baseline.
* Hx of stereotaxic brain surgery for PD.

Ages: 39 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 1999-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay S. Schneider, Ph.D., Principal Investigator — Parkinson's Disease Research Unit, Thomas Jefferson University
Locations (1):
- Parkinson's Disease Research Unit, Thomas Jefferson University, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy-seven PD patients were recruited from all across the US for this single center, double-blind, delayed start trial of GM1. Seventeen subjects participated in the comparison group. Enrollment for the study began Nov 1999 and was completed in Jan 2006. Subjects were seen at the Parkinson's Disease Research Unit at Thomas Jefferson University.
Groups:
- Early-Start Group: Phase I: Thirty nine subjects were randomized to receive GM1 for 24 weeks.
- Delayed-Start Group: Phase I: Thiry eight subjects were randomized to receive placebo for 24 weeks.
- Comparison Group: This group of PD patients who received standard of care were followed for one to two years to provide comparative information about natural disease progression. This group was not statistically compared to the treatment groups since this group was not randomized.
Period: Overall Study
Arm/Group | Early-Start Group | Delayed-Start Group | Comparison Group
Started | 39 | 38 | 17
Completed | 29 | 31 | 16
Not Completed | 10 | 7 | 1
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 1
Not completed — Protocol Violation | 2 | 2 | 0
Not completed — Unrelated Medical Problem | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early-Start Group | Delayed-Start Group | Comparison Group | Total
Number analyzed (Participants) | 39 | 38 | 17 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 29 | 9 | 65
  >=65 years | 12 | 9 | 8 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 59.7 (8.4) | 57.7 (8.7) | 61.1 (11.8) | 59.5 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 3 | 22
  Male | 29 | 29 | 14 | 72
Region of Enrollment [Number; unit: participants]
  United States | 39 | 38 | 17 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) (Part III) Motor Score From Baseline to Week 24 Assessed Off Medication.
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) (Part III) motor scores assess 14 symptoms some of which separately assess symptoms in different body parts (e.g. right arm, left arm, right leg, left leg) and each symptom is rated on a scale from 0 (normal) to 4 (severe). The minimum total score possible is 0 and the maximum total score possible is 108. Each subject was independently rated by two observers at each study visit and a mean score was calculated for analysis.
Time Frame: Baseline to Week 24
Population: Analysis was per protocol. Two subjects randomized to the Early-Start group withdrew from the study shortly after starting. The comparison group was not compared statistically to the treatment group since they were not randomized.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Groups:
- Early-Start Group: Group that was randomized to receive GM1 ganglioside 24 weeks
- Delayed-Start Group: Group that was randomized to receive placebo for 24 weeks
Arm/Group | Early-Start Group | Delayed-Start Group
Number analyzed (Participants) | 37 | 38
Scores on a scale | -3.57 (.503) | 1.85 (.497)
Statistical Analysis 1: Comparison: Early-Start Group vs Delayed-Start Group; The null hypothesis for Phase I was that at week 24, there is no difference between UPDRS motor scores in placebo vs. GM1-treated subjects; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Primary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) (Part III) Motor Scores From Baseline to Week 120 Assessed Off Medication.
Description: as for outcome 1
Time Frame: Baseline to Week 120
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Early-Start Group | Delayed-Start Group
Number analyzed (Participants) | 37 | 38
Scores on a scale | -1.80 (1.117) | 1.53 (1.092)
Statistical Analysis 1: Comparison: Early-Start Group vs Delayed-Start Group; The null hypothesis for Phase II is that long-term use of GM1 does not affect the progression of PD symptoms and that there is no benefit to early start of GM1 use; Test type: Superiority or Other; p = 0.0368, t-test, 2 sided

3. Post Hoc Outcome: Estimated Change in Points Per Week on Unified Parkinson's Disease Rating Scale (UPDRS) Motor Score Assessed Off Medication
Description: Unified Parkinson's Disease Rating Scale (UPDRS) A four part scale used to assess the severity of Parkinson's disease symptoms. Part I contains questions concerning the patient's mentation, behavior and mood. Part II asks questions about the patient's ability to perform activities of daily living. Part III is the motor examination of the patient's symptoms ranging in scores from 0 to 4 with 0 equaling either normal or absence of symptoms. The minimum score on this section is 0 and the maximum is 108. Part IV asks the patient questions about any complications of therapy they have experienced within the past week. However, for this study the total UPDRS included Parts I, II, and III. A higher the score on the scale indicates more severe symptoms.
Time Frame: Week 6 to Week 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Early-Start Group | Delayed-Start Group
Number analyzed (Participants) | 37 | 38
Scores on a scale | 0.04 (0.03) | 0.08 (0.03)
Statistical Analysis 1: Comparison: Early-Start Group; Test type: Superiority or Other; p = 0.1903, estimate of slope of change over time; random intercept model and a variance components covariance structure
Statistical Analysis 2: Comparison: Delayed-Start Group; Test type: Superiority or Other; p = 0.0063, estimate slope of change over time; random intercept model and a variance components covariance structure

4. Post Hoc Outcome: Estimated Rate of Change in Unified Parkinson's Disease Rating Scale (UPDRS)Motor Scores Assessed Off Medication
Time Frame: Week 36 to Week 120
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Early-Start Group | Delayed-Start Group
Number analyzed (Participants) | 37 | 38
Scores on a scale | 0.02 (0.01) | 0.04 (0.01)
Statistical Analysis 1: Comparison: Early-Start Group; Test type: Superiority or Other; p = 0.0502, estimate of slope of change over time; random intercept model and a variance components covariance structure
Statistical Analysis 2: Comparison: Delayed-Start Group; Test type: Superiority or Other; p = 0.0003, estimate slope of change over time; random intercept model and a variance components covariance structure

5. Secondary Outcome: Change From Baseline to Week 24 in Total Unified Parkinson's Disease Rating Scale (UPDRS)Score Assessed Off Medication
Description: The total Unified Parkinson's Disease Rating Scale (UPDRS) score is derived from Part I (Mentation, Behavior and Mood), Part II (Activities of Daily Living) and Part III (Motor Examination). Part I assesses 4 functions; Part II assesses 13 activities of daily living; Part III assesses 14 motor symptoms. Each item is rated on a scale from 0 (normal) to 4 (severe). The minimum total score possible is 0 and the maximum total score possible is 176. Each subject was independently rated by two observers at each study visit and a mean score was calculated for analysis.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Early-Start Group | Delayed-Start Group
Number analyzed (Participants) | 37 | 38
Scores on a scale | -5.31 (0.84) | 1.88 (0.83)
Statistical Analysis 1: Comparison: Early-Start Group vs Delayed-Start Group; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Change in Total UPDRS Score From Baseline to Week 120 Assessed Off Medication
Description: as for outcome 5
Time Frame: Baseline to Week 120
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Early-Start Group | Delayed-Start Group
Number analyzed (Participants) | 37 | 38
Scores on a scale | -1.01 (1.764) | 3.56 (1.726)
Statistical Analysis 1: Comparison: Early-Start Group vs Delayed-Start Group; Test type: Superiority or Other; p = 0.1310, t-test, 2 sided

7. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) (Part III) Motor Score From Baseline to Week 24 Assessed Off Medication.
Description: as for outcome 1
Time Frame: Baseline to Week 24
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Comparison Group
Number analyzed (Participants) | 17
Scores on a scale | 2.28 (0.866)
Statistical Analysis 1: Comparison: Comparison Group; Analysis was paired sample t-test on change from baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

8. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) (Part III) Motor Score From Baseline to Week 48 Assessed Off Medication.
Description: as for outcome 1
Time Frame: Baseline to Week 48
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Comparison Group
Number analyzed (Participants) | 16
Scores on a scale | 4.41 (1.434)
Statistical Analysis 1: Comparison: Comparison Group; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

9. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) (Part III) Motor Score From Baseline to Week 72 Assessed Off Medication.
Description: as for outcome 1
Time Frame: Baseline to Week 72
Population: Number of subjects enrolled at this time point.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Comparison Group
Number analyzed (Participants) | 10
Scores on a scale | 5.95 (1.220)
Statistical Analysis 1: Comparison: Comparison Group; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

10. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) (Part III) Motor Score From Baseline to Week 96 Assessed Off Medication.
Description: as for outcome 1
Time Frame: Baseline to Week 96
Population: Number of subjects enrolled at this time point.
Measure: Mean (Standard Error); unit: Scores on scale
Arm/Group | Comparison Group
Number analyzed (Participants) | 8
Scores on scale | 7.81 (2.014)
Statistical Analysis 1: Comparison: Comparison Group; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 2 and a half years beginning at baseline.
Arm/Group | Early-Start Group | Delayed-Start Group | Comparison Group
Serious Adverse Events (participants affected / at risk) | 2/39 | 1/38 | 0/17
Other Adverse Events (participants affected / at risk) | 39/39 | 38/38 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early-Start Group (N=39) | Delayed-Start Group (N=38) | Comparison Group (N=17)
Severe weakness L>R BLC LE's (General disorders) | 1 (1) | 0 (0) | 0 (0)
CT Scan showed an Ulcerating Mass Fungating in Stomach (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Increase frequency of dyskinesias (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Uncontrollable shaking (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Laproscopic Removal of Stomal Tumor in Stomach (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early-Start Group (N=39) | Delayed-Start Group (N=38) | Comparison Group (N=17)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 20 (20) | 32 (32) | 0 (0)
Injection site erythema (General disorders) | 18 (18) | 22 (22) | 0 (0)
Injection site nodule (General disorders) | 11 (11) | 17 (17) | 0 (0)
Injection site haemorrhage (General disorders) | 8 (8) | 12 (12) | 0 (0)
Injection site haematoma (General disorders) | 9 (9) | 8 (8) | 0 (0)
Injection site pruritus (General disorders) | 11 (11) | 6 (6) | 0 (0)
Injection site swelling (General disorders) | 3 (3) | 5 (5) | 0 (0)
Injection site urticaria (General disorders) | 5 (5) | 3 (3) | 0 (0)
Fatigue (General disorders) | 3 (3) | 4 (4) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 3 (3) | 0 (0)
Injection site induration (General disorders) | 2 (2) | 2 (2) | 0 (0)
Oedema (General disorders) | 2 (2) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 2 (2) | 0 (0)
Feeling abnormal (General disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site exfoliation (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Blood cholesterol increased (Investigations) | 7 (7) | 4 (4) | 0 (0)
Blood triglycerides increased (Investigations) | 6 (6) | 5 (5) | 0 (0)
Eosinophil count increased (Investigations) | 3 (3) | 3 (3) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Crystal urine present (Investigations) | 1 (1) | 2 (2) | 0 (0)
Alkaline amniotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Aspartate amnotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 9 (9) | 5 (5) | 0 (0)
Tremor (Nervous system disorders) | 5 (5) | 5 (5) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 4 (4) | 0 (0)
Dyskinesia (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Freezing phenomenon (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Vivid dreams (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No